CLINICAL TRIAL: NCT00426491
Title: Misoprostol for the Medical Management of Non-Viable First Trimester Pregnancies
Brief Title: Misoprostol for Non-Viable Pregnancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Jasmine Han, MD, Madigan Army Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 99077
Record Dates: First submitted 2007-01-22; First posted 2007-01-24 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-02

CONDITIONS: Abortifacient Agents, Nonsteroidal; Abortion, Incomplete; Misoprostol; Pregnancy
MeSH Terms: conditions — Abortion, Incomplete | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Four 200 ug tablets of Misoprostol
  Interventions: Drug: Misoprostol
- B (Placebo Comparator)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 400 ug Misoprostol or placebo will be placed in the posterior fornix of the vagina using a speculum under the direct visualization of the provider.
  Other Names: Cytotec

SUMMARY:
The purpose of this study is to examine the effectiveness of Misoprostol (Cytotec; GD Searle and Co., Chicago, IL) for the management of non-viable first trimester pregnancies. Specifically, Misoprostol (15-S-15-methyl PGE1) will be compared to a placebo with expectant management in who have documented non-viable gestations. We will examine the following outcome variables: time to resolution, number of patients requiring dilation and curettage, change in hematocrit, cost to the institution, patient satisfaction, and reported side effects.

DETAILED DESCRIPTION:
Patients presenting to the OB/GYN clinic with a nonviable gestation, diagnosis documented by endovaginal ultrasound will be enrolled. Ultrasonic findings will be verified by two of the resident staff from the obstetrics and gynecology department of Madigan Army Medical Center. Patients consenting will be directed to the OB/GYN clinic for evaluation, exam, and counseling and to watch the video giving explanation of purpose of the study and the planned procedure, but also expected side effects and possible complications. Patients will be randomized into two groups: study group receiving Misoprostol per vagina and the control group receiving a placebo per vagina. Subjects will be issued an envelope and go to the pharmacy to pick up their study medication, blinded to them and the provider. They will also be given Motrin and Phenergan to help alleviate undesired side effects. Four 200 ug tablets of Misoprostol or placebo will be placed in the posterior fornix of the vagina using a speculum under the direct visualization of the provider. Patients will return in 24 hours for re-examination. If no evidence of an intrauterine pregnancy remains, patients will be informed that their miscarriage was complete, given precautions and asked to make an appointment for follow-up in 4 weeks in addition to weekly visits to the lab for quantitative BHCG. All patients will be followed until the quantitative BHCG has fallen zero to ensure resolution of the pregnancy event.

Patients with evidence of a gestational sac will be given a second dose of Misoprostol or a D&C if they choose to withdraw from the study or a surgical intervention if it is deemed clinically indicated by the attending staff. Again, subjects will be given appropriate counseling and precautions and asked to follow up in an additional 24 hours for re-evaluation. Surveys will be given at each visit and follow up to evaluate patient satisfaction and also to query for unintended side effects and complications.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients with nonviable pregnancy document by ultrasound
* Gestation at or less than 13 weeks by ultrasound measurements
* Clinically stable as determined by provider
* Afebrile
* Hematocrit > 30
* Over 18 years of age

Exclusion Criteria:

* History of allergy to, or intolerance of, misoprostol
* Refusal to abstain from intercourse for 72 hours
* Significant vaginal bleeding (> 2 pad/hr)
* History of inflammatory bowel disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 1999-03; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
time to resolution | 24hrs, and then weekly, after insertion
percentage requiring dilation and curettage | 24hrs, and then weekly, after insertion
failure to expel products of conception | 24hrs, and then weekly, after insertion
change in hematocrit | 24hrs, and then weekly, after insertion
side effects | 24hrs, and then weekly, after insertion
BHCG level | 24hrs, and then weekly, after insertion

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Han, MD, Principal Investigator — Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States